CLINICAL TRIAL: NCT02894593
Title: Alcohol-free Essential Oils Containing Mouthrinse Efficacy on 3-day Supragingival Plaque Regrowth: a Randomized Crossover Clinical Trial
Brief Title: Alcohol-free Essential Oils Containing Mouthrinse Efficacy on 3-day Supragingival Plaque Regrowth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Adjunct Professor, University of L'Aquila
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RCT_001_16
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Gingivitis; Periodontitis
Keywords: Antiplaque agents; chemical plaque control; oral hygiene; essential oils; alcohol; mouthwash
MeSH Terms: conditions — Gingivitis; Periodontitis | interventions — Ethanol; Listerine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- alcohol essential oils mouthwash (Other): All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Other: alcohol essential oils mouthwash
- 0.20% chlorhexidine mouthwash (Active Comparator): All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Other: 0.20% chlorhexidine mouthwash
- Placebo (Placebo Comparator): All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Other: Placebo
- alcohol free essential oils mouthwash (Experimental): All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Other: alcohol free essential oils mouthwash

INTERVENTIONS:
Other: alcohol free essential oils mouthwash — All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: Listerine Zero, Johnson & Johnson Consumer Inc.
  Arms: alcohol free essential oils mouthwash
Other: alcohol essential oils mouthwash — All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: Listerine, Johnson & Johnson Consumer Inc.
  Arms: alcohol essential oils mouthwash
Other: 0.20% chlorhexidine mouthwash — All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: Meridol Chlorhexidine 0.20, GABA International AG
  Arms: 0.20% chlorhexidine mouthwash
Other: Placebo — All subjects were instructed to rinse twice a day, in the morning and in the evening, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the antiplaque effects of an alcohol-free essential-oil containing mouthrinse - Listerine Zero (LZ) and an alcohol-based essential oils (EO+) mouthwash compared to a positive control of 0.20% chlorhexidine (CHX) mouthwash, and a negative control of a placebo solution (saline), using an in vivo plaque regrowth model of 3 days.

DETAILED DESCRIPTION:
Plaque is a biofilm of microorganisms responsible for the development of caries and periodontal disease. The daily removal of supragingival dental plaque represents a major factor in the prevention of caries, gingivitis and periodontitis. Plaque control is largely obtained by daily effective tooth brushing and inter-dental cleaning, but in some cases plaque removal can be improved by adding the use of a mouthwash.

An effective action of chemical formulation (especially antiseptics) to control plaque and gingivitis levels has been proved.

Most mouthwashes contain an alcohol (especially ethanol) in order to act as a carrier agent for active essential oils to penetrate the plaque, and to give the subject a "clean mouth sensation".

The alcohol content of mouthwashes, besides having antiseptic properties, serves the purpose of breaking down or dissolving active principles, in addition to that of preserving the formula components, although such content does not directly contribute to effective biofilm and gingivitis control.

However, there are some contraindications in the use of alcohol-based mouthwashes, like the use by infants, pregnant women, alcohol addicts and patients with mucosal injuries. There are also some undesirable effects, like burning or sore sensation, or a painful sensation for patients with existing soft tissue injuries, or a perception of dryness in the mouth.

In order to avoid the use of alcohol-based mouthwashes in particular conditions, scientific interest is becoming more widespread in introducing a mouthrinse with strong anti-plaque qualities and no alcoholic ingredients.

One of these product is the alcohol-free essential oil mouthwash Listerine Zero (LZ), that has little documentation with regard to its anti-plaque effects.

The aim of this study was to evaluate the antiplaque effects of an alcohol-free essential oil mouthwash (Listerine Zero, LZ) and a alcohol-based essential oil mouthwash (EO+), compared to a positive control of a 0.2% chlorhexidine mouthwash (CHX), and a negative control of a placebo solution (saline), using an in vivo plaque regrowth model of 3 days.

The study was designed as a double-masked, randomized, crossover clinical trial, involving 21 volunteers to compare four different mouthwashes, using a 3-day plaque regrowth model. After receiving thorough professional prophylaxis at baseline, over the next 3 days, each volunteer refrained from all oral hygiene measures and performed two daily rinses with 15 ml of the test mouthwashes. EO+ was compared to LZ. CHX rinse served as a positive control, and a placebo solution as a negative control. At the end of each experimental period, plaque index (PI) was assessed, and a panelists completed through a visual analogue scale (VAS) questionnaire evaluating the organoleptic properties of each product. Each subject underwent a 14-day washout period, and then there was another allocation.

ELIGIBILITY:
Inclusion Criteria:

* dentition with ≥ 20 evaluable teeth (minimum of five teeth per quadrant)
* age between 20 and 50 years old

Exclusion Criteria:

* oral lesions
* severe periodontal problems (probing depth ≥5 mm or attachment loss >2 mm)
* removable prostheses or orthodontic bands/ or appliances
* Subjects allergic to several mouthrinse

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Dental plaque regrowth by clinical plaque index | 3 days
  all of the volunteers were examined with an erythrosine solution, and the plaque in both groups was recorded at six sites per tooth using the Quigley and Hein index , as modified by Turesky et al. and further modified by Lobene et al.

CONTACTS AND LOCATIONS:
Overall Officials: GIUSEPPE MARZO, DMD, Study Chair — University of L'Aquila
Locations (1):
- University of L'Aquila, Division of Periodontology, L’Aquila, AQ, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marchetti E, Mummolo S, Di Mattia J, Casalena F, Di Martino S, Mattei A, Marzo G. Efficacy of essential oil mouthwash with and without alcohol: a 3-day plaque accumulation model. Trials. 2011 Dec 15;12:262. doi: 10.1186/1745-6215-12-262. PMID 22171999
- [Result] Marchetti E, Casalena F, Capestro A, Tecco S, Mattei A, Marzo G. Efficacy of two mouthwashes on 3-day supragingival plaque regrowth: a randomized crossover clinical trial. Int J Dent Hyg. 2017 Feb;15(1):73-80. doi: 10.1111/idh.12185. Epub 2015 Nov 2. PMID 26522915
- [Result] Paraskevas S, Rosema NA, Versteeg P, Van der Velden U, Van der Weijden GA. Chlorine dioxide and chlorhexidine mouthrinses compared in a 3-day plaque accumulation model. J Periodontol. 2008 Aug;79(8):1395-400. doi: 10.1902/jop.2008.070630. PMID 18672988
- [Result] Charles CA, Amini P, Gallob J, Shang H, McGuire JA, Costa R. Antiplaque and antigingivitis efficacy of an alcohol-free essential-oil containing mouthrinse: a 2-week clinical trial. Am J Dent. 2012 Aug;25(4):195-8. PMID 23082381
- [Derived] Marchetti E, Tecco S, Caterini E, Casalena F, Quinzi V, Mattei A, Marzo G. Alcohol-free essential oils containing mouthrinse efficacy on three-day supragingival plaque regrowth: a randomized crossover clinical trial. Trials. 2017 Mar 31;18(1):154. doi: 10.1186/s13063-017-1901-z. PMID 28359280